CLINICAL TRIAL: NCT01075685
Title: Evaluation of an Internet-based Intervention for Hazardous Drinkers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut national de prevention et d'education pour la sante (Other Government)
Responsible Party: Guillemont, Institut national de prevention et d'education pour la sante
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Evalcoometre
Record Dates: First submitted 2010-01-06; First posted 2010-02-25 (Estimated); Results first posted 2010-11-10 (Estimated); Last update posted 2010-11-10 (Estimated); Status verified 2010-01

CONDITIONS: Hazardous Alcohol Consumption
MeSH Terms: interventions — Ethanol; Economics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Web-based alcohol programme (Experimental): Participants could log on to their account and access the programme whenever they wanted to.
  They received automated email reminders inviting them to use follow-up tools, especially the diary in order to register their alcohol intake on the previous week:
  * 4 weeks after starting the programme, so that they would take advantage of the monitoring stage in case they had not spontaneously done so.
  * 2 weeks later for 6-week follow-up.
  Interventions: Behavioral: interactive online programme to reduce alcohol consumption
- Minimum information (Placebo Comparator): Participants could log on to their account and access the programme whenever they wanted to. At 6 week follow-up they received an automated email reminder inviting them to use the diary in order to register their alcohol intake on the previous week.
  Interventions: Behavioral: Minimum information

INTERVENTIONS:
Behavioral: interactive online programme to reduce alcohol consumption — The programme includes several steps:
  * personalized feedback on alcohol consumption and related risks
  * reviewing motivations and fears regarding drinking reduction
  * analyse of drinking habits
  * reduction goal setting
  * follow-up tools (alcohol diary, craving scales, well-being scales)
  * a final screen allowing participants to monitor their progress through graphs and automatically adapted comments.
  Arms: Web-based alcohol programme
Behavioral: Minimum information — This intervention includes:
  * information about hazardous drinking
  * an alcohol diary
  Arms: Minimum information

SUMMARY:
The purpose of this study is to determine whether the investigators internet-based intervention is effective to help hazardous drinkers reducing their alcohol consumption.

ELIGIBILITY:
Inclusion Criteria:

* Alcohol Use Disorders Identification Test (AUDIT) score from 6 (female) or 7 (male) to 12

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1157 (Actual)
Dates: Start 2009-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juliette Guillemont, MS, Principal Investigator — Institut national de prevention et d'education pour la sante

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: Oct 27 to Dec 15, 2009 Recruitment was conducted via Internet.
Period: Overall Study
Arm/Group | Web-based Alcohol Programme | Minimum Information
Started | 743 | 414
Met Inclusion Criteria | 734 | 413
Completed Baseline Measures | 225 | 263
Completed | 151 | 188
Not Completed | 592 | 226
Not completed — Protocol Violation | 9 | 1
Not completed — Withdrawal by Subject | 20 | 5
Not completed — Lost to Follow-up | 563 | 220

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Web-based Alcohol Programme | Minimum Information | Total
Number analyzed (Participants) | 734 | 413 | 1147
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 718 | 408 | 1126
  >=65 years | 16 | 5 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 232 | 130 | 362
  Male | 502 | 283 | 785
AUDIT score [Mean (Standard Deviation); unit: Units on a scale] — The Alcohol Use Disorders Identification Test (AUDIT) consists of 10 questions about recent alcohol use, alcohol dependence symptoms, and alcohol-related problems. Each question has a set of responses to choose from, and each response has a score ranging from 0 to 4. All the response scores are then added, which gives the AUDIT score.
  AUDIT score ranges from 0 to 40 and is interpreted as follows:
  * 5 (female) / 6 (male) or less: low-risk drinking
  * 6 (female) / 7 (male) to 12: hazardous drinking
  * 13 or more: possible alcohol dependence.
  Units on a scale | 8.7 (1.9) | 8.8 (1.8) | 8.7 (1.8)
Weekly alcohol intake at baseline [Mean (Standard Deviation); unit: standard drinks] — Number of participants for this measure: 225 in intervention group, 263 in control group.
  The unit of "standard drink" is a drink containing 10g of pure alcohol. Participants had to report their weekly alcohol intake in a diary, in which they could choose among 21 glasses of various capacities and containing various alcoholic drinks. Each of those glasses was then converted into standard drinks.
  standard drinks | 17.5 (13.3) | 16.2 (13.2) | 16.8 (13.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Weekly Alcohol Intake
Description: The unit of "standard drink" is a drink containing 10g of pure alcohol. Participants had to report their weekly alcohol intake in a diary, in which they could choose among 21 glasses of various capacities and containing various alcoholic drinks. Each of those glasses was then converted into standard drinks.
Time Frame: baseline and 6 weeks
Population: Only participants who completed the study were included in this analysis
Measure: Mean (Standard Deviation); unit: standard drinks
Arm/Group | Web-based Alcohol Programme | Minimum Information
Number analyzed (Participants) | 151 | 188
standard drinks | -3.34 (12.19) | -1.21 (10.86)
Statistical Analysis 1: Comparison: Web-based Alcohol Programme vs Minimum Information; Test type: Superiority or Other; p = 0.0279, Type 3 tests of fixed effects

2. Secondary Outcome: Relative Change in Weekly Alcohol Intake
Description: (6 weeks minus baseline)/baseline
Time Frame: baseline and 6 weeks
Population: Participants with weekly alcohol consumption baseline at 0 were excluded from this analysis
Measure: Mean (Standard Deviation); unit: percent of baseline consumption
Arm/Group | Web-based Alcohol Programme | Minimum Information
Number analyzed (Participants) | 148 | 176
percent of baseline consumption | -0.51 (97.58) [-100 to 507.14] | 11.22 (99.89) [-100 to 692]
Statistical Analysis 1: Comparison: Web-based Alcohol Programme; Test type: Superiority or Other; p = 0.0189, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Category of Change in Weekly Alcohol Intake
Description: Category of change in weekly alcohol intake (WAI) is a 3-level categorical variable whose values are:
  * clinically significant reduction in WAI, defined as a decrease of 10% or over;
  * clinically significant increase in WAI, defined as an increase of 10% or over if WAI at baseline is positive, or any increase if WAI at baseline is 0);
  * and no clinically significant change, which includes all other cases.
Time Frame: baseline and 6 weeks
Measure: Number; unit: participants
Arm/Group | Web-based Alcohol Programme | Minimum Information
Number analyzed (Participants) | 151 | 188
participants
  significant reduction in weekly alcohol intake | 93 | 87
  no significant change in weekly alcohol intake | 7 | 13
  significant increase in weekly alcohol intake | 42 | 63
Statistical Analysis 1: Comparison: Web-based Alcohol Programme vs Minimum Information; Test type: Superiority or Other; p = 0.009, Chi-squared

4. Secondary Outcome: Change in the Number of Excessive Drinkers
Description: The number of excessive drinkers is the number of participants whose weekly alcohol intake exceeds guidelines, i.e. 21 or 14 standard drinks (male/female) per week
Time Frame: baseline and 6 weeks
Measure: Number; unit: participants
Arm/Group | Web-based Alcohol Programme | Minimum Information
Number analyzed (Participants) | 151 | 188
participants | -11 | -5
Statistical Analysis 1: Comparison: Web-based Alcohol Programme vs Minimum Information; Test type: Superiority or Other; p = 0.082, Chi-squared

ADVERSE EVENTS:
Description: Neither serious nor other adverse events were assessed.
Arm/Group | Web-based Alcohol Programme | Minimum Information
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
High rate of loss to follow-up lead to small number of subjects analyzed. Some participants were lost to follow-up even before completing baseline measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes